CLINICAL TRIAL: NCT04922073
Title: Practical Usability of EGFR Mutation Detection in ctDNA From Resectable NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: GENECAST Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Jhingook Kim, MD, Professor, Samsung Medical Center
Other Study IDs: 2021-04-150
Record Dates: First submitted 2021-05-26; First posted 2021-06-10 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating tumor DNA in plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the practical usability of EGFR mutation detection in ctDNA from early NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical stage IB to IIIA Non-small Cell Lung Cancer
* Patients with resectable lung cancer
* One of followings: 1) Never-smokers or ex-smokers who quit 10 years ago, 2) Female 3) Subsolid nodule in chest CT 4) Biopsy-proven adenocarcinoma

Exclusion Criteria:

* Patients with metastatic lung cancer (Stage IIIB-IV)
* Patients who underwent chemotherapy or radiotherapy
* Patients with other malignancies

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with clinical stage IB to IIIA Non-small Cell Lung Cancer
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Performance of the EGFR assay | Immediately before the surgery
  ADPS EGFR Mutation Test using plasma sample from clinical stage IB-IIIA NSCLC patients (reference: EGFR assay in tissue specimen)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea